CLINICAL TRIAL: NCT06516211
Title: A Candidate - Predicate Comparison and Lay User-HCP Comparison Study of the Clara(TM) Multi-Level Urine hCG Pregnancy Test
Brief Title: Predicate and Lay User-HCP Comparison Study of a Multi-Level Urine hCG Pregnancy Test
Status: Not yet recruiting | Type: Observational
Sponsor: Conceptra Biosciences, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: CCT-101.001
Record Dates: First submitted 2024-06-10; First posted 2024-07-23 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Pregnancy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Lay User
  Interventions: Device: Clara Pregnancy Test
- HCP Predicate Device
  Interventions: Device: Clara Pregnancy Test; Device: Professional Marketed Pregnancy Test

INTERVENTIONS:
Device: Clara Pregnancy Test — Multi-Level Pregnancy Test
Device: Professional Marketed Pregnancy Test — Early Pregnancy Test
  Groups: HCP Predicate Device

SUMMARY:
Study volunteers will be required to conduct a home pregnancy test (HPT) at the trial center and provide a sample of urine from the same void for further testing.

Volunteers will then complete a product usage questionnaire and leaflet comprehension questionnaire at site.

DETAILED DESCRIPTION:
Eligible volunteers will be recruited into the study and provide informed consent.

Volunteers will then test their urine sample with the investigational HPT according to the device Instructions For Use, and their results will be recorded. A sample of urine from the same void will be obtained for further testing by the healthcare provider (HCP) study technicians.

The HCP technician will then test the volunteer's sample with a second investigational HPT, a professional use pregnancy test and a HPT, the results of which will be used to provide the volunteer with her pregnancy test result. During technician testing, the volunteer will complete the device usability and leaflet comprehension questionnaires.

True pregnancy status will be determined by laboratory tests and clinical information.

ELIGIBILITY:
Inclusion Criteria:

* Females (persons assigned female at birth and not sterile) willing and able to provide written consent to Study participation
* Able to read and write in English or Spanish

Exclusion criteria:

* Persons employed in a healthcare or laboratory setting and/or with professional experience who conduct point of care urine tests
* Previous or current enrollment in a Clara™ Study
* Visually or otherwise impaired to a degree they are not able to readily read and follow instructions, or visualize the faint pink lines.
* Unwilling or unable to provide at least 12mls of urine specimen and any urine testing they are expected to receive as a part of their non-Study related care.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Persons assigned female at birth and not sterile
Study Population: Females over the age of 18, who are capable of becoming pregnant.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2025-09-30 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Lay-Professional Comparison | 1 day
  Demonstration of agreement of pregnancy test reading. The agreement between lay participant test results and those of a technician testing the same urine sample.

SECONDARY OUTCOMES:
Predicate Comparison | 1 day
  Demonstration of agreement of pregnancy test reading. The agreement between the predicate device and investigational device test results performed by a technician testing the same urine sample.

CONTACTS AND LOCATIONS:
Locations (1):
- FPA Women's Health, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No